CLINICAL TRIAL: NCT05309434
Title: Effects of CPR Coaching on Leader's Performance During Simulated Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EESOA11
Record Dates: First submitted 2022-03-22; First posted 2022-04-04 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Leadership
MeSH Terms: interventions — Doulas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group with standing coach (Experimental): The team performs the simulated CPR with the coach standing next to the defibrillator
  Interventions: Behavioral: Coach
- study group with mobile coach (Experimental): The team performs the simulated CPR with the coach free to move around the simulation room
  Interventions: Behavioral: Coach
- control group without coach (No Intervention): The team performs the simulated CPR without the coach

INTERVENTIONS:
Behavioral: Coach — The coach coordinates the initiation of CPR, communicates feedback device data to assist those performing compressions, communicates average targets for compressions and ventilations and coordinates operations to achieve those values, and communicates with the team to reduce pauses in compressions.
  Arms: Study group with standing coach; study group with mobile coach

SUMMARY:
Previous studies reported that the introduction of the role of the CPR Coach in resuscitation teams led to an increase in the adherence of CPR to AHA guidelines by the team.

To date, the interaction between the CPR Coach and the Team Leader during the performance of CPR remains poorly studied.

In this study, the investigators aim to evaluate whether the interaction between the CPR Coach and the Team Leader brings real benefits to the cognitive engagement of the latter and therefore whether or not his leadership and the overall performance of the team is affected.

DETAILED DESCRIPTION:
In this study, 60 trainees will be divided into 10 teams of 6 participants each, which include two CPR providers, a team leader, a nurse actor, a defibrillator actor with (study groups A and B) or without (control group, C) a coach.

Each team will perform a standardized 10-minute cardiopulmonary resuscitation (CPR) simulation on a standardized Trauma Hal mannequin (Gaumard Scientific) with a Combat Application Tourniquet (CAT Resources, Rock Hill, SC)/SUSIE simulator(Gaumard Scientific, Miami, FL) with a CPR Feedback device. All participants assigned the role of the coach will receive standardized training as described by Cheng et al, 2018.

Study group A will run the simulation with the CPR coach figure standing next to the defibrillator; study group B will run the simulation with the CPR coach free to move around the scenario; control group C will run the simulation without the CPR coach. During the simulations, an experienced facilitator and a simulation technician will be present to conduct and oversee the progress of the activities.

All activities of all teams will be recorded with cameras and microphones. At the end of each simulation, there will be a debriefing conducted by an expert facilitator to make the simulation experience complete but will not be considered in the study.

All recorded videos will be viewed by 4 experts who will score the leader's performance and the team's performance. The leader's performance will be evaluated by using the Resuscitation Team Leader Evaluation Scale (RTLE) (Grant et al,2012). The Team's overall performance will be evaluated by the Clinical Performance Toll (CPT)(Donoghue et al, 2010).

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia trainees
* Emergency medicine trainees

Exclusion Criteria:

* none

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
Team leader performance | 30 minutes
  Evaluation of team leader's performance by using the Resuscitation Team Leader Evaluation Scale (RTLE) (0=not performed or not observed; 1= performed but ineffectively, incompletely, or inconsistently; 2=performed adequately most of the time; 3= performed well consistently). High scores are the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Azienda Universitaria Ospedaliera, Padua, Italy

REFERENCES:
- [Background] Grant EC, Grant VJ, Bhanji F, Duff JP, Cheng A, Lockyer JM. The development and assessment of an evaluation tool for pediatric resident competence in leading simulated pediatric resuscitations. Resuscitation. 2012 Jul;83(7):887-93. doi: 10.1016/j.resuscitation.2012.01.015. Epub 2012 Jan 28. PMID 22286047
- [Background] Cheng A, Duff JP, Kessler D, Tofil NM, Davidson J, Lin Y, Chatfield J, Brown LL, Hunt EA; International Network for Simulation-based Pediatric Innovation Research and Education (INSPIRE) CPR. Optimizing CPR performance with CPR coaching for pediatric cardiac arrest: A randomized simulation-based clinical trial. Resuscitation. 2018 Nov;132:33-40. doi: 10.1016/j.resuscitation.2018.08.021. Epub 2018 Aug 24. PMID 30149088
- [Background] Donoghue A, Nishisaki A, Sutton R, Hales R, Boulet J. Reliability and validity of a scoring instrument for clinical performance during Pediatric Advanced Life Support simulation scenarios. Resuscitation. 2010 Mar;81(3):331-6. doi: 10.1016/j.resuscitation.2009.11.011. Epub 2010 Jan 4. PMID 20047787